CLINICAL TRIAL: NCT02072070
Title: A Placebo Controlled, Double-blind, Randomized, Parallel-group, Multi-center Phase III Study to Determine the Efficacy and Safety of TissueGene-C in Patients With Degenerative Arthritis
Brief Title: Efficacy and Safety Study of TissueGene-C to Degenerative Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS-TGC-01-3
Record Dates: First submitted 2014-02-17; First posted 2014-02-26 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Degenerative Arthritis
Keywords: chondrocyte cells, Osteoarthritis, gene therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TissueGene-C (Experimental): Single intra-articular injection to the damaged knee joint at a dose of 1.8 x 10^7 cells
  Interventions: Biological: TissueGene-C
- Placebo (Placebo Comparator): Single intra-articular injection to the damaged knee joint
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: TissueGene-C — TissueGene-C at 1.8 x 10^7 cells
  Arms: TissueGene-C
Drug: Placebo — Placebo control(Normal Saline)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether TissueGene-C, an allogeneic human chondrocytes expressing Transforming Growth Factor(TGF)-b1, is effective and safe in patients with degenerative arthritis.

DETAILED DESCRIPTION:
TissueGene-C is a biological new drug which consists of normal chondrocyte cells and transduced chondrocyte cells that express growth factor to modify osteoarthritis symptom for long term period.

During the Phase 3 clinical trial , we will compare TissueGene-C to placebo in 26, 52 weeks trial with 156 outpatients who have osteoarthritis. The outpatients are randomized to TissueGene-C or placebo in 1:1 ratio, and they will be monitored and recorded in terms of alleviating symptoms, sports activities, function of the knee, and the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 19 years of age
2. Patients diagnosed with degenerative arthritis
3. Patients with IKDC(Knee Documentation Committee subjective score) score of 60 or below
4. Patients with 100 mm VAS(Visual Analog Scale) score of 40 or above
5. With Grade 3 osteoarthritis as determined by the radiographic criteria of Kellgren and Lawrence
6. With an International Cartilage Repair Society(ICRS) Grade III or IV cartilage damage in the major lesions, as confirmed through an MRI scan
7. With a Body Mass Index(BMI) of higher than18.5 and lower than 30
8. Patients who satisfies the clinical/radiational criteria by the American College of Rheumatology (ACR) guidelines, and applies to one of the following.

   * Older than 50
   * Morning stiffness for less than 30 minutes
   * Crepitus and Osteophytes
9. With major lesions concentrated in one section of the knee, and with the major lesions considered the main cause of the clinical symptoms
10. With no alleviation of the symptoms even after at least three months of non-surgical treatment
11. Healthy, with no major findings from the physical examination, hematology, serum chemistry, and urine tests, and no significant medical history
12. Agreed to use an effective contraceptive method during the study period
13. Voluntarily agreed to participate in this study, and signed the informed consent form

Exclusion Criteria:

1. Showed clinically significant hematology, serum chemistry, and urine test results at the screening visit
2. Regarding inclusion criteria 6. following patients should not be included

   * patients with a major lesion of ICRS grade 4 which is larger than 6cm2(for patient with ICRS grade 4)
   * patients with a major lesion of ICRS grade 3 which is larger than 6cm2(for patient without a ICRS grade 4),
3. Patient who had skin disease around target knee
4. patients who have a positive skin reaction to CS-10
5. Patients who had been administered with drugs such as oriental medicine, glucosamine and chondroitin within 14 days of baseline visit
6. Patients taking steroidal anti-inflammatory medications within 14 days of baseline visit
7. Patients with severe pain in other areas that could effect the diagnosis of the symptoms of the
8. History of surgery like arthroendoscopy within the past 6 months on the target knee
9. Patients who had been administered with immunosuppressants, including antirheumatic drugs (including methotrexate or antimetabolite), within the past 3 months
10. Patients who had been treated with physical therapy or herbal remedy (acupuncture, heat etc.) within 2 weeks of baseline visit
11. History of injection within the past 3 months on the target knee
12. Pregnant or breastfeeding female
13. With another joint disease apart from degenerative arthritis (e.g., systemic rheumatic inflammatory disease associated with the knee or chondrocalcinosis, hemachromatosis, inflammatory arthritis, necrosis of the trochanter, Paget's disease adjacent to a joint in the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's disease in the knee joint, villonodular synovitis, synovial chondromas)
14. With an infectious disease, including HIV or hepatitis
15. With any of the following clinically significant diseases:

    * heart disease (e.g., myocardial infarction, arrhythmia, other serious heart diseases, coronary artery bypass graft)
    * kidney disease (e.g., chronic renal failure, glomerulonephritis)
    * liver disease (e.g., liver cirrhosis, fatty liver, acute or chronic liver disease)
    * endocrine disease (e.g., hyperthyroidism, hypothyroidism, thyroiditis, diabetes insipidus, Cushing's disease)
    * insulin-dependent diabetes mellitus
    * medical history of past or current malignant tumor
    * In particular, the tumors that TissueGene-C may aggravate can be screened using the following tests:

      * Leukemia (White Blood Cell level in the hematology)
      * Osteochondroma, Chondromas, Chondroblastoma, Chondromyxoid fibroma, Chondrosarcoma (Alkaline phosphatase level in the hematology)
16. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
17. Patients who administered the TissueGene-C from past clinical trial
18. Considered inappropriate by the investigator for participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in IKDC scores | Week 0 and 52
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)
Changes in 100 mm VAS scores | Week 0 and 52
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Changes in WOMAC scores | Wekk 0, 26, 39 and 52
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
Changes in KOOS scores | Week 0, 26, 39 and 52
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Changes in MRI scan | Week 0, 26 and 52
  Comparison of pre-procedure MRI scans to those obtained at pre-dosing and at months 6 and 12 following dosing by an independent radiographic reviewer.
Changes in Joint Space Width by an independent radiographic reviewer. | Week 0, 26 and 52
Level of Biomarkers in blood and urine. | Week 0, 26, 39 and 52
Proportion of Patients Use of Rescue Medication. | Week 4, 12, 26, 39 and 52
Changes in IKDC scores | Week 0, 26 and 39
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)
Changes in 100 mm VAS scores | Week 0, 26 and 39
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Gu Kim, MD, PhD, Principal Investigator — Inje University; Su Hee Kyung, MD, PhD, Principal Investigator — Kyungpook National University Hospital; Chul Won Ha, MD, PhD, Principal Investigator — Samsung Medical Center; Myung Chul Lee, MD, PhD, Study Chair — Seoul National University Hospital; Yong In, MD, PhD, Principal Investigator — The Catholic University of Korea Seoul ST. Mary's Hospita; Seong Il Bin, MD, PhD, Principal Investigator — Asan Medical Center; Seong Do Cho, MD, PhD, Principal Investigator — Ulsan University Hospital; Jae Doo Yoo, MD, PhD, Principal Investigator — Ewha Womans University Mokdong; Myung Gu Kim, MD, PhD, Principal Investigator — Inha University Hospital; Ju Hong Lee, MD, PhD, Principal Investigator — Chonbuk National University Hospital; Ui Seong Choi, MD, PhD, Principal Investigator — Chungbuk National University Hospital; Chung Hyeok Choi, MD, PhD, Principal Investigator — Hanyang University
Locations (12):
- South Korea (12):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National Univ. Hospital, Daegu
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Inje University Seoul Paik Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Chen L, Huang FL, Tang Q, Zhao ZK, Ye ZY, Liang JH. Targeted therapy for knee osteoarthritis: From basic to clinics. Medicine (Baltimore). 2025 Aug 15;104(33):e43686. doi: 10.1097/MD.0000000000043686. PMID 40826764
- [Derived] Kim MK, Ha CW, In Y, Cho SD, Choi ES, Ha JK, Lee JH, Yoo JD, Bin SI, Choi CH, Kyung HS, Lee MC. A Multicenter, Double-Blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of a Cell and Gene Therapy in Knee Osteoarthritis Patients. Hum Gene Ther Clin Dev. 2018 Mar;29(1):48-59. doi: 10.1089/humc.2017.249. PMID 29641281